CLINICAL TRIAL: NCT03298932
Title: 2D Strain of Right Ventricle in Peroperative Cardiac Surgery : Evaluation of Early Signs of RV Dysfunction
Brief Title: 2D Strain of Right Ventricle in Peroperative of Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9597
Record Dates: First submitted 2016-10-11; First posted 2017-10-02 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2016-10

CONDITIONS: Aortic Valve Disorder
Keywords: Transesophageal echography; Perioperative cardiac surgery; Aortic valve replacement; 2D strain of right ventricle
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Aortic valve surgery — Aortic valve surgery

SUMMARY:
Evaluation of the right ventricle (RV) deformation (strain) with 2D speckle tracking technics obtained by echocardiographies (TEE) in peroperative period of cardiac surgery .

TEE is performed for each patient of cardiac surgery during the operation time .

This new evaluation parameter of RV could be a good tool to assess the early RV dysfunction after cardiac surgery.

DETAILED DESCRIPTION:
Monitoring of 2D strain of right ventricle free wall by TEE in perioperative of cardiac surgery :

In preoperative time After sternotomy After surgery Inclusions of patients elected for aortic valve surgery without coronary diseases or previous RV dysfunction.

Comparison with others echocardiographic parameters of RV evaluation Association with right ventricle insufficiency after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient eligible for aortic valve surgery

Exclusion criteria:

* previous right ventricle dysfunction
* severe coronary disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible for aortic valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
2D strain modification of right ventricle after cardiac surgery | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine CULAS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hôpital Arnaud de Villeneuve réanimation, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided